CLINICAL TRIAL: NCT01378429
Title: A 6-Week Randomized, Double-blind, Placebo-controlled, Parallel Group, Safety Study of the Potential Inhibitory Effects of Ciclesonide Nasal Aerosol on the Hypothalamic-Pituitary-Adrenal (HPA) Axis in Subjects 6-11 Years With Perennial Allergic Rhinitis (PAR)
Brief Title: Safety Study of the Potential Inhibitory Effects of Ciclesonide Nasal Aerosol on the Hypothalamic-Pituitary-Adrenal Axis in Subjects 6-11 Years With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060-308
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Perennial Allergic Rhinitis; PAR
Keywords: Perennial Allergic Rhinitis; PAR
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ciclesonide nasal aerosol (Experimental): ciclesonide nasal aerosol (74 mcg)
  Interventions: Drug: ciclesonide nasal aerosol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ciclesonide nasal aerosol — ciclesonide nasal aerosol (74 mcg)
  Arms: ciclesonide nasal aerosol
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group, safety study of the effects of ciclesonide nasal aerosol (74 mcg) on the HPA axis when administered once daily to male and premenarchal female subjects 6 to 11 years of age with a diagnosis of PAR.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group, safety study of the effects of ciclesonide nasal aerosol (74 mcg) on the HPA axis when administered once daily to male and premenarchal female subjects 6 to 11 years of age with a diagnosis of PAR.

The study requires that subjects be domiciled during two 24- to 36-hour time periods for sample collection for serum and urinary free cortisol measurements, as well as PK evaluations (single [predose] time point during the first domiciled period, and 24-hour sampling during the second domiciled period).

ELIGIBILITY:
Inclusion Criteria:

* Gives written informed consent (parent/legal guardian) and assent (when appropriate, from the child), including privacy authorization as well as adherence to concomitant medication withholding periods, prior to participation.
* Is a male or premenarchal female 6 to 11 years old and ≥ 20 kg at the screening visit.
* Is in general good health (defined as the absence of any clinically relevant abnormalities as determined by the investigator) based on screening physical examination and medical history.
* Has a history of PAR to a relevant perennial allergen (house dust mites, cockroaches, molds, animal dander) for a minimum of one year immediately preceding the study screening visit. The PAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past and require treatment throughout the entire study period.
* Has a demonstrated sensitivity to at least one allergen known to induce PAR (house dust mites, cockroaches, molds, and animal dander) based on a documented result with a standard skin-prick test either within one year prior to the screening visit or performed at the screening visit. A positive test is defined as a wheal diameter at least 3 mm larger than the negative control wheal for the skin-prick test. The subject's positive allergen test must be consistent with the medical history of of PAR, and the allergen must be present in the subject's environment throughout the study.

Exclusion Criteria:

* Has a history of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations; recent nasal biopsy; nasal trauma; or nasal ulcers or perforations. Surgery and atrophic rhinitis or rhinitis medicamentosa are not permitted within the 120 days prior to the screening visit.
* Has evidence of infection, significant anatomic abnormality, ulceration of the mucosa, blood in the nose, or any other clinically relevant finding on nasal examination at the screening visit.
* Has nasal jewelry.
* Has participated in any investigational drug trial within the 30 days preceding the screening visit or is planning participation in another investigational drug trial at any time during this trial.
* Has a known hypersensitivity to any corticosteroid or any of the excipients in the formulation of ciclesonide.
* Has a history of a respiratory infection or disorder, including but not limited to bronchitis, pneumonia, influenza, and severe acute respiratory syndrome (SARS), within the 14 days preceding the screening visit.
* Has a history of adrenal insufficiency.
* Has active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta-agonists and any controller drugs (eg, theophylline, leukotriene antagonists); intermittent use (≤ 3 uses per week) of inhaled short-acting beta-agonists is acceptable. Use of short-acting beta-agonists for exercise-induced bronchospasm will be allowed.
* Is expecting to use any disallowed concomitant medications during the treatment period.
* Is, in the investigator's judgment, having a seasonal exacerbation at the time of the screening visit.
* Is planning initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the screening visit and use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
* Has nonvaccinated exposure to or active infection with chickenpox or measles within the 21 days preceding the screening visit.
* Initiates pimecrolimus cream 1% or greater or tacrolimus ointment 0.03% or greater during the study period or plans a dose escalation during the study period. However, initiation of these creams/ointments 30 days or more prior to screening and use of a stable (maintenance) dose during the study period may be considered for inclusion.
* Has experienced significant blood loss within 60 days or loss of plasma within 72 hours prior to the screening visit or intends to undergo elective surgery within 30 days following end of study.
* Is a child or immediate relative of any clinical investigator or site personnel, even those who are not directly involved in this study.
* Resides in the same household as another subject who is participating in this study at the same time.
* Has any of the following conditions that are judged by the investigator to be clinically significant and/or to affect the subject's ability to participate in the clinical trial:

  * impaired hepatic function
  * history of ocular disturbances, eg, glaucoma or posterior subcapsular cataracts or herpes simplex
  * any systemic infection
  * hematological (including anemia), hepatic, renal, endocrine disease
  * gastrointestinal disease
  * malignancy (excluding basal cell carcinoma)
  * current neuropsychological condition with or without drug therapy. Any behavioral condition that could affect subject's ability to accurately report symptoms to the caregiver such as developmental delay, attention deficit disorder, and autism.
* Has any condition that, in the judgment of the investigator, would preclude the subject from completing the protocol with capture of the assessments as written.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - West Coast Clinical Trials, Costa Mesa, California
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Sneeze, Wheeze, & Itch Associates, LLC, Normal, Illinois
  - Clinical Research Institute, Plymouth, Minnesota
  - Western Sky Medical Research, El Paso, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvania Research Associates, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Started | 42 | 47
Completed | 41 | 47
Not Completed | 1 | 0
Not completed — Noncompliance with study drug | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo nasal aerosol administered once daily (1 actuation per nostril)
- Ciclesonide Nasal Aerosol (74 mcg): Ciclesonide nasal aerosol 74 mcg administered once daily (1 actuation of 37 mcg per nostril)
- Total: Total of all reporting groups
Arm/Group | Placebo | Ciclesonide Nasal Aerosol (74 mcg) | Total
Number analyzed (Participants) | 42 | 47 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (1.74) | 8.6 (1.65) | 8.9 (1.70)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 47 | 89
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 20 | 25 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 29 | 35 | 64
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 17 | 32
  Not Hispanic or Latino | 27 | 30 | 57
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 47 | 89

OUTCOME MEASURES:

1. Primary Outcome: The Change in Serum Cortisol Area Under the Curve (AUC) From Time 0 to 24 Hours (0-24), Calculated Using a Trapezoidal Rule, From Baseline to the End of the 6 Week Treatment Period
Description: Area under the concentration-time curve from time 0 to 24 hours [AUC(0-24h)]. Timepoints at which data were collected: 0, 2, 4, 8, 12, 16, and 24 at week 0 and 6.
Time Frame: Week 0 and 6
Population: The Per Protocol (PP) population consisted of all ITT subjects who had sufficient blood sample collection at Visit 4/BL and Visit 7/End of Week 6 for serum cortisol measurements, completed the study on treatment medication and had no important protocol deviations (IPDs).
Measure: Least Squares Mean (Standard Error); unit: mcg•hour/dL
Groups:
- Ciclesonide Nasal Aerosol: Ciclesonide nasal aerosol 74 mcg administered once daily (1 actuation of 37 mcg per nostril)
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 39 | 46
mcg•hour/dL | 5.9 (5.6) | -1.7 (5.2)
Statistical Analysis 1: Comparison: Placebo vs Ciclesonide Nasal Aerosol; 35 subjects per arm would have ≥90% power to demonstrate that the upper bound of a two-sided 95% confidence interval (equivalent to the upper bound of a one-sided 97.5% confidence interval) of the difference of placebo minus ciclesonide nasal aerosol would be less than 20% of the baseline value of 175 mcg•h/dL or a noninferiority limit of 35 mcg•h/dL assuming a SD of 40 and a one-sided α of 0.025. A total of 40 subjects will be randomly assigned to ensure 35 subjects complete the study per arm; Test type: Non-Inferiority or Equivalence — 35 subjects per arm would have ≥90% power to demonstrate that the upper bound of a two-sided 95% confidence interval (equivalent to the upper bound of a one-sided 97.5% confidence interval) of the difference of placebo minus ciclesonide nasal aerosol would be less than 20% of the baseline value of 175 mcg•h/dL or a noninferiority limit of 35 mcg•h/dL assuming a SD of 40 and a one-sided α of 0.025. A total of 40 subjects will be randomly assigned to ensure 35 subjects complete the study per arm; ANCOVA — <0.025 for a one-sided test; LS Mean Difference = 7.6, 95% CI 2-sided [-7.4 to 22.6] — Difference is calculated as Placebo - Ciclesonide

2. Secondary Outcome: Change From Baseline in Urinary Free Cortisol-Corrected for Urine Creatinine
Time Frame: weeks 0-6
Population: The PP population. Subjects with either missing baseline data or post dose data, or both were not included in the analysis
Measure: Least Squares Mean (Standard Error); unit: mcg/g
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 39 | 45
mcg/g | 1.4 (2.9) | 3.3 (2.7)

3. Secondary Outcome: Change From Baseline in Urinary Free Cortisol-Uncorrected for Urine Creatinine
Time Frame: weeks 0-6
Population: The PP population consisted of all ITT subjects who had sufficient blood sample collection at Visit 4/BL and Visit 7/End of Week 6 for serum cortisol measurements, completed the study on treatment medication and had no IPDs.
Measure: Least Squares Mean (Standard Error); unit: mcg/g
Groups:
- Placebo: Placebo nasal aerosol administered once daily (1 actuation per nostril) for 6 weeks
- Ciclesonide Nasal Aerosol: Ciclesonide nasal aerosol 74 mcg administered once daily (1 actuation of 37 mcg per nostril) for 6 weeks
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 39 | 45
mcg/g | 0.5 (1.9) | 1.2 (1.8)

4. Secondary Outcome: Number of Subjects Experiencing AEs
Time Frame: weeks 0-6
Population: Intent-to-treat (ITT) Population: All randomized subjects who received at least 1 dose of double blind study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 42 | 47
participants
  Any AE | 19 | 20
  Potentially related AE | 6 | 4
  Nasal (local) AEs | 6 | 5
  Discontinued study drug due to an AE | 0 | 0
  Severe AE | 1 | 0
  Serious AE | 0 | 0
  Death | 0 | 0

5. Secondary Outcome: Percentage of Subjects Experiencing AEs
Time Frame: weeks 0-6
Population: Intent-to-treat (ITT) Population: All randomized subjects who received at least 1 dose of double blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 42 | 47
percentage of participants
  Any AE | 45.2 | 42.6
  Potentially related AE | 14.3 | 8.5
  Nasal (local) AEs | 14.3 | 10.6
  Discontinued study drug due to an AE | 0 | 0
  Severe AE | 2.4 | 0
  Serious AE | 0 | 0
  Death | 0 | 0

6. Secondary Outcome: Number of Subjects Experiencing Nasal AEs, Including Epistaxis, Nasal Ulceration, and Nasal Perforation.
Description: Local Treatment-Emergent Adverse Events (ITT Population)
Time Frame: weeks 0-6
Population: Intent-to-treat (ITT) Population: All randomized subjects who received at least 1 dose of double blind study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 42 | 47
participants
  Overall | 6 | 5
  Epistaxis | 2 | 1
  Mucosal erosion | 1 | 0
  Nasal discomfort | 1 | 1
  Postnasal drip | 0 | 1
  Rhinitis | 1 | 0
  Rhinorrhea | 0 | 1
  Traumatic hemorrhage | 1 | 0
  Upper respiratory tract infection | 0 | 1
  Viral upper respiratory tract infection | 2 | 0

7. Secondary Outcome: Percentage of Subjects Experiencing Nasal AEs, Including Epistaxis, Nasal Ulceration, and Nasal Perforation.
Description: Local Treatment-Emergent Adverse Events (ITT Population)
Time Frame: weeks 0-6
Population: Intent-to-treat (ITT) Population: All randomized subjects who received at least 1 dose of double blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 42 | 47
percentage of participants
  Overall | 14.3 | 10.6
  Epistaxis | 4.8 | 2.1
  Mucosal erosion | 2.4 | 0
  Nasal discomfort | 2.4 | 2.1
  Postnasal drip | 0 | 2.1
  Rhinitis | 2.4 | 0
  Rhinorrhea | 0 | 2.1
  Traumatic hemorrhage | 2.4 | 0
  Upper respiratory tract infection | 0 | 2.1
  Viral upper respiratory tract infection | 4.8 | 0

8. Secondary Outcome: AUC(0-24h)
Description: Area under the concentration-time curve from time 0 to 24 hours. Collected at 0, 30 min, 60 min, 90 min, 2 hours (h), 4 h, 8 h, 12 h, 16 h, and 24h after dosing.
Time Frame: Week 6
Population: PK Population: Subjects in the ITT population who completed the study on treatment medication and had assayed serum concentrations of ciclesonide and/or des ciclesonide. Descriptive statistics were presented for serum drug/metabolite concentrations and evaluable pharmacokinetic parameters.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 47
ng*hr/mL
  Ciclesonide serum concentration | 0.072 (0.261)
  Des-ciclesonide serum concentration | 0.261 (0.139)

9. Secondary Outcome: Maximum Observed Concentration
Description: Cmax (ng/mL) (PK Population)
Time Frame: Week 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 47
ng/mL
  Ciclesonide serum concentration | 0.012 (0.0009)
  Des-ciclesonide serum concentration | 0.029 (0.0169)

10. Secondary Outcome: Time to the Occurrence of Cmax
Description: tmax (hour) (PK Population)
Time Frame: Week 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 47
Hour
  Ciclesonide serum concentration | 1.146 (0.700)
  Des-ciclesonide serum concentration | 2.200 (1.330)

11. Secondary Outcome: Terminal Half Life (t1/2)
Description: Terminal half-life (t1/2) (hour)
Time Frame: Weeks 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 47
Hour
  Ciclesonide serum concentration | 8.194 (12.448)
  Des-ciclesonide serum concentration | 11.727 (5.864)

12. Secondary Outcome: Apparent Clearance of the Drug (CL/F)
Description: CL/F liter per hour (L/hour) is the apparent clearance of the drug
Time Frame: Week 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 47
L/hour
  Ciclesonide serum concentration | 1222.4 (573.99)
  Des-ciclesonide serum concentration | 317.8 (190.49)

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Vz/F Liters (L) is the apparent volume of distribution
Time Frame: Week 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 47
L
  Ciclesonide serum concentration | 34831.4 (35986.86)
  Des-ciclesonide serum concentration | 6151.3 (7999.78)

14. Secondary Outcome: Ratio (Percentage) of the Number of Correct Advances of the Dose Indicator to the Number of Expected Advances Based on Subject Self-report of Study Medication Administration Plus Extra Non-nasal Actuations
Time Frame: weeks 0-6
Population: Intent-to-treat (ITT) Population: All randomized subjects who received at least 1 dose of double blind study medication.
Measure: Mean (Standard Deviation); unit: percentage of number of correct advances
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 42 | 47
percentage of number of correct advances | 101.75 (9.647) | 100.73 (11.637)

15. Secondary Outcome: Number of Devices With Actuation Consistency, Where Actuation Consistency is Defined as a Dose Indicator Count Within ± 20% of the Subject Self-report of Study Medication Administration
Time Frame: weeks 0-6
Population: Intent-to-treat (ITT) Population: All randomized subjects who received at least 1 dose of double blind study medication.
Measure: Number; unit: Devices
Units Other Than Participants: Devices
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 42 | 47
Number analyzed (Devices) | 123 | 141
Devices | 112 | 126

16. Secondary Outcome: Percentage of Devices With Actuation Consistency, Where Actuation Consistency is Defined as a Dose Indicator Count Within ± 20% of the Subject Self-report of Study Medication Administration
Time Frame: weeks 0-6
Population: Intent-to-treat (ITT) Population: All randomized subjects who received at least 1 dose of double blind study medication.
Measure: Number; unit: percentage of devices
Units Other Than Participants: Devices
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 42 | 47
Number analyzed (Devices) | 123 | 141
percentage of devices | 91.1 | 89.4

17. Secondary Outcome: Change From Baseline in Averaged Daily Subject-reported AM and PM Reflective TNSS Averaged Over the 6 Weeks of Double-blind Treatment
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent 1 = mild 2 = moderate 3 = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the six week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement
Time Frame: weeks 0-6
Population: Intent-to-treat (ITT) Population: All randomized subjects who received at least 1 dose of double blind study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Number analyzed (Participants) | 42 | 47
units on a scale | -0.7 (1.65) | -1.5 (2.04)

ADVERSE EVENTS:
Time Frame: 0-6 weeks
Arm/Group | Placebo | Ciclesonide Nasal Aerosol
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/47
Other Adverse Events (participants affected / at risk) | 5/42 | 3/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | Ciclesonide Nasal Aerosol (N=47)
Headache (Nervous system disorders) | 1 (3) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.